CLINICAL TRIAL: NCT01447823
Title: Observational Field Study of Acute Esophageal Food Bolus Impaction by Mean Esophageal Manometry and 24h-pH-monitoring
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: KEK-ZH Nr 2011-0192
Record Dates: First submitted 2011-09-27; First posted 2011-10-06 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Esophageal Motility Disorders
Keywords: Oesophageal bolus obstruction; Gastroscopy; phmetry
MeSH Terms: conditions — Esophageal Motility Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of this study is to evaluate standard investigations performed in patients with bolus impaction in a prospective observational field study. In bolus impaction, ingested food boluses have to be endoscopically removed. Oesophageal narrowing by scar tissue caused by reflux disease or motility disorders are possible causes of bolus impaction. How common these causes are has up to date never been investigated. The discovery of eosinophilic oesophagitis has broadened differential diagnosis of bolus impaction. Currently high resolution oesophageal manometry and 24-hour pHmetry are performed in addition to endoscopy in the assessment of bolus impaction at the University Hospital Zurich.

The collection of these examination results is the aim of this prospective unrandomised observational field study to assess weather the currently applied procedures are valid to diagnose the cause of impaction to find optimal therapy for each patient.

DETAILED DESCRIPTION:
The key function of the esophagus ist (i) the immediate transport of the food bolus from the mouth to the stomach and (ii) to inhibit reflux from the stomach back to the esophagus.

Motility disorders of the esophagus lead to an impaired bolus transport and/or reflux of stomach content to the esophagus, and may cause symptoms such as (obstructive) dysphagia, chest pain, heart burn and/or regurgitation.

Acute esophageal food impaction is a common acute condition of the upper GI tract that usually needs immediate medical attention. The food bolus, e.g. a peace of red meat or similar is blocked within the tubular part of the esophagus, e.g. proximal to the esophagogastric junction and neither passes spontaneously into the stomach nor can be regurgitated actively. In this case it usually requires upper endoscopy for endoscopic removal of the food bolus.

Possible causes of food impaction are (i) structural obstruction within the esophagus such as a Schatzki's ring, an esophageal web, a peptic stenosis secondary to gastroesophageal reflux disease, or more rarely esophageal carcinoma [1, 2]; (ii) functional causes of obstruction are mainly Achalasia or Esophageal Esophagitis (EE). In Achalasia a idiopathic neurodegenerative destruction of the inhibitory neurons of the esophagus leads to a failure of the lower esophageal sphincter to relax and an impaired esophageal peristalsis. Patients usually present with a history of progressive dysphagia and regurgitation of undigested food, but rarely a food impaction can occur [3]. Eosinophilic Esophagitis is a idiopathic disorder in which eosinophilic infiltration of the mucosal wall leads to an impaired esophageal motility, which usually causes dysphagia, retrosternal pain or food bolus impaction.[3] Its etiology remains unknown but several studies suggest an allergic response to food and allergens. Previously believed to be a rather rare disease and therefore rare cause for bolus impaction, eosinophilic esophagitis has emerged as one of the most common causes for food impaction and dysphagia in general [4]. The increase in prevalence is not entirely clear; besides better recognition by gastroenterologists and pathologists there seems to be a true increase in incidence, probably due to an increased incidence of allergic diseases [5]. Its diagnosis is difficult due to other causes of eosinophilic infiltrate such as gastroesophageal reflux disease or eosinophilic gastroenteritis[3].

The reason for an impaired motility in EE is unknown, although several hypothetic mechanisms are discussed [6]: (i) increased contraction of fibroblast secondary to presence of eosinophilic granulocytes, (ii) axonal necrosis secondary to eosinophilic degradation (iii) binding of eosinophil derived MBP (major basic protein) to muscarinic acetylcholine receptors leading to increased contraction.

The true prevalence of eosinophilic esophagitis in patients with food impaction remains unknown. Desai et al evaluated 31 patients with acute bolus impaction of which more than 50% had an increased count of intraesophageal eosinophils per high power field [4]. However, the true share of EE remains unclear. Especially the amount of patients with eosinophilic infiltrate due to gastroesophageal reflux is not defined (half of all patients had PPI before endoscopy).

The current clinical standard of care for patients with food bolus impaction at the Division of Gastroenterology at the University Hospital Zurich includes

1. endoscopy to i) remove the food bolus; ii) take esophageal, gastric and duodenal biopsies to assess histological abnormalities and iii) assess structural causes for obstruction;
2. a high resolution esophageal manometry (HRM) to assess esophageal motility;
3. an ambulatory intraesophageal pH-monitoring to asses esophageal acid exposure and
4. venous blood sampling to assess eosinophilic count in peripheral blood.

These procedures are considered to be both i) necessary as well as ii) sufficient and accurate to elucidate the true cause of bolus impaction [3]. Our aim is now to objectify this standard procedure of care in an open, prospective, observational, unrandomized field study. It is important to mention that all procedures have been and are indicated in this situation as current standard procedure of care to assess patients with bolus impaction; they should be performed whether the patient is included in our field study or not. Therefore participation in the study does not lead to any additional diagnostic or therapeutic procedures/interventions

ELIGIBILITY:
Inclusion criteria:

* Patients with acute esophageal bolus impaction coming to the emergency unit of the University Hospital Zurich needing emergency endoscopy for bolus removal
* Age > 18 years
* Informed consent

Exclusion criteria:

* Age under 18 years
* Inability to understand the informed consent form

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing upper endoscopy for removal of a food bolus are asked to sign the standard clinical informed consent form for interventional endoscopy of the Division of Gastroenterology at the University Hospital Zurich. After Diagnosis of food impaction has been made, the food bolus has been removed and the endoscopy has been completed, the patient will be informed of the Diagnosis and the standard procedure of care (High resolution manometry, pH-monitoring, blood sampling) will be explained, and an appointment for these procedures will be given (1-4days thereafter).
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2011-08; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich; Michael Fried, Professor, MD, Principal Investigator — University Hospital Zurich, Division of Gastroenterology and Hepatology
Locations (1):
- University Hospital Zurich, Gastroenterology and Hepatology, Zurich, Switzerland